CLINICAL TRIAL: NCT03702244
Title: Prospective Randomized Trial of the Optimal Evaluation of Cardiac Symptoms and Revascularization
Brief Title: The PRECISE Protocol: Prospective Randomized Trial of the Optimal Evaluation of Cardiac Symptoms and Revascularization
Acronym: PRECISE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: HeartFlow, Inc. (Industry)
Collaborators: Duke Clinical Research Institute (Other); Cardiovascular Research Foundation, New York (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: CP-907-001-A
Record Dates: First submitted 2018-10-03; First posted 2018-10-11 (Actual); Results first posted 2023-12-29 (Actual); Last update posted 2023-12-29 (Actual); Status verified 2023-10

CONDITIONS: Coronary Artery Disease
Keywords: suspected coronary artery disease
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Intervention Model Description: Participants who meet all inclusion criteria and none of the exclusion criteria will be randomized in a ratio of 1:1 within a clinical center to either a precision evaluation strategy or usual care using an interactive web or voice-based system (IXRS). Randomization will be stratified by intended first test if randomized to usual care and by classification as minimal vs. elevated risk by the minimal risk model. The randomization scheme within a clinical center will be carried out by the method of random permuted block design with variable block size
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- Usual Care (No Intervention): For participants randomized to usual care, the participant's care team will select the specific noninvasive stress test (exercise electrocardiogram, stress nuclear imaging [including PET], stress MR, or stress echocardiogram); OR invasive test: (direct to diagnostic catheterization).
- Precision evaluation (Other): Participants randomized to a precision strategy will be assigned to either guideline-recommended care without immediately planned testing (low risk) or cCTA with selective FFRct (elevated risk) using a risk tool based on pretest clinical characteristics derived from the PROMISE trial and validated in SCOT-HEART trial. Participants assigned to guideline-recommended care without planned testing will be treated with preventive and antianginal medical treatment per guideline recommendations and clinical judgment and followed without testing.
  Interventions: Diagnostic Test: cCTA with selective FFRct

INTERVENTIONS:
Diagnostic Test: cCTA with selective FFRct — PRECISE will evaluate whether a precision evaluation strategy that combines contemporary risk stratification using the PROMISE Risk Tool with functional and anatomic non-invasive evaluation with cCTA with selective FFRct can improve outcomes over usual care in stable chest pain patients while safely deferring further testing in low-risk patients and reducing cost overall
  Arms: Precision evaluation

SUMMARY:
The study will be a prospective, pragmatic, randomized clinical trial of the comparative effectiveness of diagnostic evaluation strategies for stable CAD, to be performed in outpatient settings, including primary care and cardiology practices.

DETAILED DESCRIPTION:
Objective was to test a modified initial cCTA strategy (PS) designed to improve clinical efficiency vs usual testing (UT). Patients from 65 North American and European sites with stable symptoms of suspected coronary artery disease (CAD) and no prior testing were randomly assigned 1:1 to precision strategy PS or UT. PS incorporated the Prospective Multicenter Imaging Study for the Evaluation of Chest Pain (PROMISE) minimal risk score to quantitatively select minimal-risk participants for deferred testing, assigning all others to cCTA with selective CT-derived fractional flow reserve (FFR-CT). UT included site-selected stress testing or catheterization. Site clinicians determined subsequent care.

ELIGIBILITY:
Inclusion criteria (all must be present):

1. Age ≥18 years
2. Stable typical or atypical symptoms suggesting possible significant coronary artery disease (CAD) with further non-emergent testing or elective catheterization recommended to evaluate the presence of suspected significant CAD. Stable chest pain (or equivalent) includes those who have fully been ruled out for Acute Coronary Syndrome (ACS) and for whom elective testing is recommended, regardless of the venue in which they are seen.
3. If prior CV testing has occurred, it must have been performed greater than one year prior to randomization, and the following must be met:

   1. cCTA or invasive coronary angiography (ICA) with stenosis < 50%
   2. Quantified coronary artery calcium (CAC) < 100 AG
4. Safe performance of cCTA:

   1. Creatinine clearance ≥45 ml/min per most recent measurement within 90 days
   2. For a female participant of childbearing potential (those who have not been surgically sterilized or are not postmenopausal), a pregnancy test must be performed with negative results known within 7 days prior to randomization
5. Willingness to comply with all aspects of the protocol, including adherence to the assigned strategy and follow-up visits
6. Ability to provide written informed consent

Exclusion criteria (all must be absent):

1. Acute chest pain (in patients who have not been ruled out for ACS)
2. Unstable clinical status
3. Noninvasive or invasive CV testing for CAD within 1 year. CV testing for CAD refers to any stress tests, invasive coronary angiography (ICA) and cCTA (including calcium scoring) only.

   a. Resting ECG, resting echocardiogram and resting CMR (MRI) are not exclusionary regardless of when were performed
4. Lifetime history of known obstructive CAD (prior myocardial infarction, CABG or PCI, stenosis ≥50%), known EF ≤40% or other moderate to severe valvular or congenital cardiac disease
5. Contraindications to cCTA including but not limited to creatinine clearance (GFR) <45 ml/min as per most recent measurement taken within 90 days
6. Exceeds the site's weight or size limit for cCTA or cardiac catheterization
7. Any condition leading to possible inability to comply with the protocol procedures or follow-up
8. Any condition that might interfere with the study procedures or follow-up
9. Enrolled in an investigational trial that involves a non-approved cardiac drug or device which has not reached its primary endpoint
10. Life expectancy less than 2 years due to non-cardiovascular comorbidities

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2103 (Actual)
Dates: Start 2018-11-27 (Actual); Primary Completion 2022-05-20 (Actual); Study Completion 2022-05-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pamela S Douglas, Principal Investigator — Duke University
Locations (1):
- Participating site, Lake Charles, Louisiana, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Chew DS, Mark DB, Li Y, Nanna MG, Kelsey MD, Daniels MR, Davidson-Ray L, Baloch KN, Rogers C, Patel MR, Anstrom KJ, Curzen N, Vemulapalli S, Douglas PS; PRECISE Investigators. Economic Outcomes With Precision Diagnostic Testing Versus Usual Testing in Stable Chest Pain: Results From the PRECISE Randomized Trial. Circ Cardiovasc Qual Outcomes. 2025 Feb;18(2):e011008. doi: 10.1161/CIRCOUTCOMES.123.011008. Epub 2025 Feb 3. PMID 39895495
- [Derived] Mark DB, Li Y, Nanna MG, Kelsey MD, Daniels MR, Rogers C, Patel MR, Baloch KN, Chow BJW, Anstrom KJ, Vemulapalli S, Weir-McCall JR, Stone GW, Chew DS, Douglas PS; PRECISE Investigators. Quality of Life Outcomes With a Risk-Based Precision Testing Strategy Versus Usual Testing in Stable Patients With Suspected Coronary Disease: Results From the PRECISE Randomized Trial. Circ Cardiovasc Qual Outcomes. 2025 Feb;18(2):e011414. doi: 10.1161/CIRCOUTCOMES.124.011414. Epub 2025 Feb 3. PMID 39895494
- [Derived] Udelson JE, Kelsey MD, Nanna MG, Fordyce CB, Yow E, Clare RM, Mark DB, Patel MR, Rogers C, Curzen N, Pontone G, Maurovich-Horvat P, De Bruyne B, Greenwood JP, Marinescu V, Leipsic J, Stone GW, Ben-Yehuda O, Berry C, Hogan SE, Redfors B, Ali ZA, Byrne RA, Kramer CM, Yeh RW, Martinez B, Mullen S, Huey W, Anstrom KJ, Al-Khalidi HR, Chiswell K, Vemulapalli S, Douglas PS; PRECISE Investigators. Deferred Testing in Stable Outpatients With Suspected Coronary Artery Disease: A Prespecified Secondary Analysis of the PRECISE Randomized Clinical Trial. JAMA Cardiol. 2023 Oct 1;8(10):915-924. doi: 10.1001/jamacardio.2023.2614. PMID 37610768
- [Derived] Douglas PS, Nanna MG, Kelsey MD, Yow E, Mark DB, Patel MR, Rogers C, Udelson JE, Fordyce CB, Curzen N, Pontone G, Maurovich-Horvat P, De Bruyne B, Greenwood JP, Marinescu V, Leipsic J, Stone GW, Ben-Yehuda O, Berry C, Hogan SE, Redfors B, Ali ZA, Byrne RA, Kramer CM, Yeh RW, Martinez B, Mullen S, Huey W, Anstrom KJ, Al-Khalidi HR, Vemulapalli S; PRECISE Investigators. Comparison of an Initial Risk-Based Testing Strategy vs Usual Testing in Stable Symptomatic Patients With Suspected Coronary Artery Disease: The PRECISE Randomized Clinical Trial. JAMA Cardiol. 2023 Oct 1;8(10):904-914. doi: 10.1001/jamacardio.2023.2595. PMID 37610731
- [Derived] Nanna MG, Vemulapalli S, Fordyce CB, Mark DB, Patel MR, Al-Khalidi HR, Kelsey M, Martinez B, Yow E, Mullen S, Stone GW, Ben-Yehuda O, Udelson JE, Rogers C, Douglas PS. The prospective randomized trial of the optimal evaluation of cardiac symptoms and revascularization: Rationale and design of the PRECISE trial. Am Heart J. 2022 Mar;245:136-148. doi: 10.1016/j.ahj.2021.12.004. Epub 2021 Dec 23. PMID 34953768

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were randomly assigned 1:1 to precision strategy (PS) or usual testing (UT), stratified by site, intended first test if randomly assigned to UT, and minimal vs moderate-high risk using the validated PROMISE minimal risk score(PMRS).
  All PS and UT testing was performed according to local protocols, and all subsequent testing and care decisions were made locally.
Groups:
- Precision Strategy (PS): Participants in the PS group with a PROMISE minimal risk score (PMRS - validated tool) threshold value of greater than 0.46 were assigned to deferred testing. All other participants in the PS group (ie, those with a PMRS <0.46), or those with known atherosclerosis such as vascular calcification on chest CT, received cCTA with selective FFR-CT for site-read 30% to 90% stenoses.
  All testing was performed according to local protocols, and all subsequent testing and care decisions were made locally.
- Usual Testing (UT): Among participants in the UT group, site clinicians chose the initial testing modality, including exercise electrocardiogram, stress echocardiogram, stress nuclear myocardial perfusion imaging (single-photon emission CT or positron emission tomography), stress cardiovascular magnetic resonance imaging, or catheterization.
  All testing was performed according to local protocols, and all subsequent testing and care decisions were made locally.
Period: Overall Study
Arm/Group | Precision Strategy (PS) | Usual Testing (UT)
Started | 1057 | 1046
Completed | 1057 | 1046
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Precision Strategy (PS): Participants were randomly assigned 1:1 to precision strategy (PS) or usual testing (UT), stratified by site, intended first test if randomly assigned to UT, and minimal vs moderate-high risk using the validated PROMISE minimal risk score(PMRS).
  Participants in the PS group with a PROMISE minimal risk score (PMRS - validated tool) threshold value of greater than 0.46 were assigned to deferred testing. All other participants in the PS group (ie, those with a PMRS <0.46), or those with known atherosclerosis such as vascular calcification on chest CT, received cCTA with selective FFR-CT for site-read 30% to 90% stenoses.
  All PS and UT testing was performed according to local protocols, and all subsequent testing and care decisions were made locally.
- Usual Testing (UT): Participants were randomly assigned 1:1 to precision strategy (PS) or usual testing (UT), stratified by site, intended first test if randomly assigned to UT, and minimal vs moderate-high risk using the validated PROMISE minimal risk score(PMRS).
  Among participants in the UT group, site clinicians chose the initial testing modality, including exercise electrocardiogram, stress echocardiogram, stress nuclear myocardial perfusion imaging (single-photon emission CT or positron emission tomography), stress cardiovascular magnetic resonance imaging, or catheterization.
  All PS and UT testing was performed according to local protocols, and all subsequent testing and care decisions were made locally.
- Total: Total of all reporting groups
Arm/Group | Precision Strategy (PS) | Usual Testing (UT) | Total
Number analyzed (Participants) | 1057 | 1046 | 2103
Age, Continuous [Mean (Standard Deviation); unit: years] | 58.0 (11.5) | 58.9 (11.6) | 58.4 (11.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 508 | 539 | 1047
  Male | 549 | 507 | 1056
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | NA — Privacy rules precluded accessing more detail about non-white race/ethnicity. | NA — Privacy rules precluded accessing more detail about non-white race/ethnicity. | NA — Total not calculated because data are not available (NA) in one or more arms.
  Asian | NA — Privacy rules precluded accessing more detail about non-white race/ethnicity. | NA — Privacy rules precluded accessing more detail about non-white race/ethnicity. | NA — Total not calculated because data are not available (NA) in one or more arms.
  Native Hawaiian or Other Pacific Islander | NA — Privacy rules precluded accessing more detail about non-white race/ethnicity. | NA — Privacy rules precluded accessing more detail about non-white race/ethnicity. | NA — Total not calculated because data are not available (NA) in one or more arms.
  Black or African American | NA — Privacy rules precluded accessing more detail about non-white race/ethnicity. | NA — Privacy rules precluded accessing more detail about non-white race/ethnicity. | NA — Total not calculated because data are not available (NA) in one or more arms.
  White | 892 | 875 | 1767
  More than one race | NA — Privacy rules precluded accessing more detail about non-white race/ethnicity. | NA — Privacy rules precluded accessing more detail about non-white race/ethnicity. | NA — Total not calculated because data are not available (NA) in one or more arms.
  Unknown or Not Reported | NA — Privacy rules precluded accessing more detail about non-white race/ethnicity. | NA — Privacy rules precluded accessing more detail about non-white race/ethnicity. | NA — Total not calculated because data are not available (NA) in one or more arms.
Hypertension [Count of Participants; unit: Participants] — Participants were randomized to either the usual care arm or the precision evaluation arm within 14 days of screening. Major cardiac risk factors were assessed (incl. hypertension) at baseline.
  Participants | 642 | 606 | 1248
Body mass index [Mean (Standard Deviation); unit: kg/m^2] | 30.2 (6.6) | 29.9 (6.2) | 30.0 (6.4)
Diabetes [Count of Participants; unit: Participants] | 176 | 197 | 373
Dyslipidemia [Count of Participants; unit: Participants] | 668 | 681 | 1349
Family history of premature CAD [Count of Participants; unit: Participants] | 404 | 395 | 799
Peripheral arterial or cerebrovascular disease [Count of Participants; unit: Participants] | 65 | 56 | 121
Current or past tobacco use [Count of Participants; unit: Participants] | 544 | 554 | 1098
Absence of any CV risk factors [Count of Participants; unit: Participants] — The precision evaluation arm starts with the use of the PROMISE Risk Tool to categorize patient risk for CAD and events. The PROMISE Risk Tool is a validated risk model that has been shown to accurately identify chest pain patients who are unlikely to benefit from non-invasive testing (i.e. have minimal or no atherosclerosis and likely to have no events within two years). Risk was classified by a risk tool using pre-test clinical characteristics (including tobacco usage, ethnicity, and age) derived in the PROMISE trial and validated in SCOT-HEART or by the presence of non-obstructive plaque.
  Participants | 67 | 61 | 128
PROMISE minimal risk score >0.46 (minimal risk) [Count of Participants; unit: Participants] | 214 | 219 | 433
Primary presenting symptom (Chest pain) [Count of Participants; unit: Participants] | 870 | 876 | 1746
Type of angina (Typical - cardiac) [Count of Participants; unit: Participants] | 249 | 257 | 506
Type of angina (Atypical - possible cardiac) [Count of Participants; unit: Participants] | 600 | 597 | 1197

OUTCOME MEASURES:

1. Primary Outcome: Primary Composite (Number) of Deaths / MIs / Invasive Coronary Angiography Without Obstructive Disease
Description: The centrally adjudicated (by Clinical Events Committee) primary end point was a composite of clinical efficiency as a gatekeeper to invasive testing (catheterization without obstructive CAD) and safety (death, non fatal myocardial infarction [MI]) at 1 year. Invasive cardiac catheterization without obstructive coronary artery disease defined as the absence of any ≥50% stenosis or hemodynamic indication of significance (no FFR ≤0.80 or iFR≤0.89) in any major epicardial vessel including side branches ≥2 mm in diameter, as determined by core-lab adjudicated quantitative coronary angiography (QCA) or if QCA not performed, by site report. A detailed description and information on the definitions of primary endpoint component definitions is provided in the current version of the study Protocol, Statistical Analysis Plan, and the published trial design article.
Time Frame: 1 year
Population: Statistical testing for recurrent events was performed using the negative binomial methods for recurrent events. The primary endpoint of this study is estimated as time to first occurrence of any of its three following components: All-cause death; Non-fatal MI; Invasive cardiac catheterization without obstructive CAD.
Measure: Number; unit: number of events
Arm/Group | Precision Strategy (PS) | Usual Testing (UT)
Number analyzed (Participants) | 1057 | 1046
number of events
  Primary Composite End Point | 44 | 118
  Death or Nonfatal Myocardial Infarction (first event only) | 18 | 12
  Death from any cause | 5 | 7
  Nonfatal Myocardial Infarction | 13 | 5
  Invasive cardiac catheterization without Obstructive coronary disease | 27 | 107
Statistical Analysis 1: Comparison: Precision Strategy (PS) vs Usual Testing (UT); Sample size and power calculations for this study are based on the hypothesis that the precision evaluation arm is superior to the usual care arm on the time-to-first event of the composite 3-component endpoint: all-cause death, non-fatal MI, or invasive cardiac catheterization without obstructive CAD over a 12-month of follow-up. Time to event analysis will use the date of the event, including the date of catheterization at which the absence of obstructive CAD is demonstrated; Test type: Superiority — Statistical testing for recurrent events was performed using the negative binomial methods for recurrent events; p < .001, Log Rank; Hazard Ratio (HR) = 0.29, 95% CI 2-sided [0.20 to 0.41] — Hazard ratio was adjusted for age, sex, and coronary artery disease equivalent (diabetes, history of peripheral artery disease or cerebrovascular disease), and intended first test strata (invasive or noninvasive)

2. Secondary Outcome: Number of Unplanned Hospitalizations (Including Admissions With Death or MI)
Description: Urgent and unscheduled hospitalizations for cardiovascular causes include hospitalization for ischemic heart disease including myocardial infarction and unstable angina, cerebrovascular disease including stroke and TIA, heart failure, acute and/or critical limb ischemia, other thrombotic events including pulmonary embolism, arrhythmias, cardiac arrest and other clear cardiovascular causes for hospitalization that do not meet the criteria for the specific events listed here (e.g., hospitalization for acute cardiac chest pain that does not meet the criteria for MI or UA).
Time Frame: 1 year
Population: For All Cause Hospitalization only a descriptive summary will be presented.
Measure: Number; unit: number of events
Arm/Group | Precision Strategy (PS) | Usual Testing (UT)
Number analyzed (Participants) | 1057 | 1046
number of events
  Cardiovascular | 31 | 21
  For Unstable Angina | 9 | 5

3. Secondary Outcome: Number of Catheterization and Revascularization Procedures
Description: Catheterization efficiency was defined as the proportion of invasive cardiac catheterization patients who undergo revascularization (PCI or CABG) within 6 months. Revascularization may occur either percutaneously (PCI) or surgically (CABG) or as hybrid (PCI and CABG). For PCI, any intervention on a lesion in the coronary tree (including angioplasty, stenting, intravascular lithotripsy) whether successful or not will be considered a revascularization. For CABG the start of the surgical procedure (skin incision) was considered as CABG, whether the procedure was successful or not. Staged revascularization was considered as one revascularization event.
Time Frame: 1 year
Population: Additionally catheterization efficiency or cath yield is defined as the proportion of participants with an invasive coronary angiogram who underwent revascularization within 6 months of catheterization. Rates will be summarized by 2 groups.
Measure: Number; unit: number of events
Arm/Group | Precision Strategy (PS) | Usual Testing (UT)
Number analyzed (Participants) | 1057 | 1046
number of events
  Invasive catheterization | 135 | 177
  Rate of finding obstructive CAD on catheterization | 108 | 70
  Total Revascularizations | 97 | 54
  PCI | 77 | 37
  CABG | 21 | 18

4. Secondary Outcome: Number of Participants With Preventive Medication Use
Description: Lipid-lowering agents included statins, ezetimibe, PCSK9 inhibitors. Antiplatelet agents included aspirin, clopidogrel, ticagrelor, or prasugrel. Antihypertensive medications included calcium channel blockers, angiotensin-converting enzyme inhibitors, angiotensin receptor blockers, angiotensin-neprilysin inhibitor, beta blockers, nitrates, or diuretics.
Time Frame: 1 Year
Population: The number (%) will be summarized between the precision care arm and usual care arm.
Measure: Count of Participants; unit: Participants
Arm/Group | Precision Strategy (PS) | Usual Testing (UT)
Number analyzed (Participants) | 900 | 873
Participants
  Antiplatelet | 321 | 237
  Lipid-lowering | 450 | 365
  Anti-hypertensive | 504 | 455

5. Secondary Outcome: Number of Participants With Quality of Life (Angina Frequency) Assessment
Description: Overall health status was assessed briefly using the EQ-5D-5L, a standardized generic measure that can also be used to link specific health states to general population-based utilities. The EQ-5D-5L consists of two parts: (1) a descriptive assessment of five dimensions (mobility, self-care, usual activities, pain/discomfort, anxiety/depression), each of which can take one of five responses corresponding to the level of severity within each dimension, and (2) a self-rating 0- 100 "thermometer" of current health-related quality of life. The proportion of participants with frequent angina (Seattle Angina Questionnaire angina frequency score <80).
Time Frame: 1 year
Population: Angina Frequency Score at Baseline was used as reference. Not all participants fully completed the questionnaire, therefore data were collected as presented below.
Measure: Count of Participants; unit: Participants
Arm/Group | Precision Strategy (PS) | Usual Testing (UT)
Number analyzed (Participants) | 894 | 868
Participants
  More frequent angina: all participants | 141 | 140
  More frequent angina: participants with typical angina: number analyzed (Participants) | 249 | 257
  More frequent angina: participants with typical angina | 50 | 40

6. Secondary Outcome: Cumulative Radiation Exposure From All Cardiovascular Procedures (12 M), MilliSievert (mSv)
Description: The cumulative radiation exposure over the 12 months following Randomization was calculated based on each participant's exposure to radiation for cardiovascular care. If data are missing in > 80% or more of the diagnostic and procedural testing, a single fixed estimate of radiation based on the literature will be used to impute. Given high missingness in catheterization data, a fixed estimate of 6.6 mSv and 4.1 mSv was used for catheterization with and without revascularization, respectively, based on recent trial data.
Time Frame: 1 year
Population: In instances in which sufficient information required to assess actual dose is not available, data were imputed. For CCTA and nuclear imaging missing values were imputed based on distribution of data from participants. Cumulative radiation exposure from additional cardiac testing and procedures during the entire follow-up period were also collected or estimated based on accepted average exposures. Given high missingness in catheterization data, a fixed estimate of 6.6 mSv and 4.1 mSv was used.
Measure: Mean (Standard Deviation); unit: mSv
Arm/Group | Precision Strategy (PS) | Usual Testing (UT)
Number analyzed (Participants) | 1057 | 1046
mSv | 5.2 (5.4) | 4.7 (6.0)

ADVERSE EVENTS:
Time Frame: 1 year
Description: Since all trial procedures represent standard of care for the eligible study population, there are no specific safety events associated with investigative procedures in this trial. However, there are known complications from these clinically recommended tests and procedures which are outlined in sections below.
  An independent clinical event committee (CEC) was responsible for the blinded review and adjudication of the primary endpoints (Death, MI and Cath without obstructive CAD).
Groups:
- Precision Strategy (PS): Participants in the PS group with a PROMISE minimal risk score (PMRS - validated tool) threshold value of greater than 0.46 were assigned to deferred testing. All other participants in the PS group (ie, those with a PMRS <0.46), or those with known atherosclerosis such as vascular calcification on chest CT, received cCTA with selective FFR-CT for site-read 30% to 90% stenoses.
  All PS and UT testing was performed according to local protocols, and all subsequent testing and care decisions were made locally.
- Usual Testing (UT): Among participants in the UT group, site clinicians chose the initial testing modality, including exercise electrocardiogram, stress echocardiogram, stress nuclear myocardial perfusion imaging (single-photon emission CT or positron emission tomography), stress cardiovascular magnetic resonance imaging, or catheterization.
  All PS and UT testing was performed according to local protocols, and all subsequent testing and care decisions were made locally.
Arm/Group | Precision Strategy (PS) | Usual Testing (UT)
All-Cause Mortality (participants affected / at risk) | 5/1057 | 7/1046
Serious Adverse Events (participants affected / at risk) | 40/1057 | 30/1046
Other Adverse Events (participants affected / at risk) | 13/1057 | 43/1046
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Precision Strategy (PS) (N=1057) | Usual Testing (UT) (N=1046)
Myocardial Infarction (MI - non-fatal) (Cardiac disorders) | 13 (13) | 5 (5) — Acute MI was defined as having evidence of myocardial necrosis in a clinical setting consistent with myocardial ischemia. Fatal MI is excluded. The Fourth Universal Definition of MI was used.
Death from any cause (Cardiac disorders) | 5 (5) | 7 (7) — All cause death is defined as death resulting from any cause.
Unplanned CV hospitalization excluding admissions with MI or death (Cardiac disorders) | 22 (23) | 18 (18) — Unplanned cardiovascular (CV) admissions to hospital without MI or death during the same episode of care. Statistical testing for recurrent events was performed using the negative binomial methods for recurrent events.
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Precision Strategy (PS) (N=1057) | Usual Testing (UT) (N=1046)
HeartFlow Analysis (FFRCT) - Customer Support Investigations (Product Issues) | 0 (0) | 0 (0) — For post-market study, all potential FFRCT - possible device related adverse events were to be immediately reported through HeartFlow Customer Support for investigation. There were zero (0) complaints/ possible device related events.
Major test and procedural complications by test type (Injury, poisoning and procedural complications) | 4 (4) | 6 (6) — There were no specific safety events associated with investigative procedures in this trial. All complications occurring (during the cardiovascular test as per protocol) were categorized in two groups (1) Major and (2) Minor, and by test type.
Minor test and procedural complications by test type (Injury, poisoning and procedural complications) | 9 (9) | 37 (37) — There were no specific safety events associated with investigative procedures in this trial. All complications occurring (during the cardiovascular test as per protocol) were categorized in two groups (1) Major and (2) Minor, and by test type.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Confidentiality embargo was in place until primary results were published.

DOCUMENTS (2):
  • Study Protocol (2018-06-29): https://cdn.clinicaltrials.gov/large-docs/44/NCT03702244/Prot_000.pdf
  • Statistical Analysis Plan (2022-07-07): https://cdn.clinicaltrials.gov/large-docs/44/NCT03702244/SAP_001.pdf